CLINICAL TRIAL: NCT04065529
Title: Efficacite et Innocuite du Tannate de Gelatine Dans le Traitement de la Diarrhee aiguë de l'Enfant. Une Etude Randomisee, Controlee, en Double Aveugle (INDIGO)
Brief Title: Clinical Trial in Children Between 3 Months and 14 Years Old to Evaluate the Efficacy and Safety of Gelatin Tannate in the Treatment of Acute Diarrhea (INDIGO)
Acronym: INDIGO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferrer Internacional S.A. (Industry)
Collaborators: Axonal-Biostatem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E870
Record Dates: First submitted 2019-06-11; First posted 2019-08-22 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Diarrhea
Keywords: Diarrhea; gastroenterology; acute gastroenteritis; gastroenteritis; acute; gelatin; tannate
MeSH Terms: conditions — Diarrhea; Gastroenteritis | interventions — tannate gelatin; World Health Organization oral rehydration solution; ORALIT

STUDY DESIGN:
Intervention Model Description: Interventional, randomized, controlled, double blind, multicenter phase III clinical trial.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gelatin tannate (GT) (Experimental): Gelatin tannate (GT)
  Interventions: Combination Product: Gelatin tannate (GT) + oral rehydration solution (ORS) + Zinc supplementation
- Placebo (Placebo Comparator): Placebo
  Interventions: Combination Product: placebo + ORS + Zinc supplementation

INTERVENTIONS:
Combination Product: Gelatin tannate (GT) + oral rehydration solution (ORS) + Zinc supplementation — Gelatin tannate (GT) + oral rehydration solution (ORS) + Zinc supplementation
  Arms: Gelatin tannate (GT)
Combination Product: placebo + ORS + Zinc supplementation — placebo + ORS + Zinc supplementation
  Arms: Placebo

SUMMARY:
To evaluate the safety, global efficacy and rapidity of action of GT in children with acute gastroenteritis taking ORS solution.

DETAILED DESCRIPTION:
Study purpose:

To evaluate the safety, global efficacy and rapidity of action of GT in children with acute gastroenteritis taking ORS solution.

Study centers/ settings: The recruitment will take place in public health facilities in Senegal.

Proposed site is the Niakhar Center IRD BP 1386 Hann Mariste, Dakar-Senegal) with the health center of Niakhar as satellite site. More sites can be opened at the discretion of the Sponsor if required

Study design and type:

Interventional, randomized, controlled, double blind, multicenter phase III clinical trial.

Test product/arms:

Gelatin tannate (GT) + oral rehydration solution (ORS) + Zinc supplementation versus (vs.) placebo + ORS + Zinc supplementation.

Investigational Product: GELATIN TANNATE (GT):

* Children below 3 years of age: One sachet every 6 hours
* Children from 3 to 14 years of age: 2 sachets every 6 hours. All patients will take ORS solution according to 2014 European recommendations, and Zinc supplementation.

Reference Product:

Placebo. The dose regimen and mode of administration will be similar as the investigational product.

Number of patients planned:

150 patients, randomized in 1:1 basis (75 in each arm).

Inclusion criteria:

Children eligible for the trial must fulfil ALL of the following criteria:

* AGE defined as a change in stool consistency to loose or liquid form (according to the Bristol Stool Form (BSF) scale ≥ 6 or, the Brussels Infant and Toddler Stool Scale (BITSS) =4 in the case of infants ≤ 3 years (see Annex 1) and/or an increase in the frequency of evacuations (typically ≥3 in 24 h),
* AGE lasting between 1 day and 2 days;
* Children from 3 months old
* Children up to 14 years old;
* Written informed consent form signed by parents or legal guardians must be provided to caregivers.
* Subject willing and able to comply with study restrictions and willing to return to the health center and to perform the follow-up evaluation as specified in the protocol.

Non-inclusion criteria: In order to participate in this study, all subjects must meet NONE of the following exclusion criteria:

* Use of antibiotics, diosmectite, probiotics, racecadotril, loperamide or zinc (including zinc containing ORS) within a week prior to enrolment
* Chronic diarrheal gastrointestinal disease (eg, inflammatory bowel diseases, cystic fibrosis, coeliac disease, food allergy)
* Immunodeficiencies
* Signs of malnutrition according to the opinion of the investigator (weight/height under 3rd z score as per World Health Organization [WHO] Child Growth Standards)
* Subject who previously entered in a clinical study within the past 30 days.
* Pregnancy and suspected Pregnancy

Study duration: 7 days including 5 days of treatment; follow up at Day 7.

Study outcomes:

Primary outcome:

The primary outcome will be the duration of diarrhea, defined as the time between start of diarrhea and the normalization of stool consistency according to the BSF or BITSS (in BSF scale, =3 or =4; in BITSS, =2), or/and the time until the normalization of the number of stools (compared with the period before the onset of diarrhea), and the presence of normal stools for 48 h.

A subgroup analysis will be performed with patients for whom the cause of the diarrhea is not parasitic.

Secondary outcomes:

* Stool Decrease Index (SDI)
* Time resolution of diarrhea from start of treatment
* Need for intravenous rehydration
* Number of watery stools per day
* Vomiting
* Weight gain
* Recurrence of diarrhea (48 h after intervention)
* Severity of diarrhea according to Vesikari scale
* Use of concomitant medications.
* Adverse events (AEs)

Expected results:

Significant decrease of duration of diarrhea with the Gelatin Tannate plus ORS plus zinc than placebo+ ORS +zinc

ELIGIBILITY:
Inclusion Criteria:

* AGE defined as a change in stool consistency to loose or liquid form (according to the Bristol Stool Form (BSF) scale ≥ 6 or, the Brussels Infant and Toddler Stool Scale (BITSS) =4 in the case of infants ≤ 3 years (see Annex 1) and/or an increase in the frequency of evacuations (typically ≥3 in 24 h),
* AGE lasting between 1 day and 2 days;
* Children from 3 months old
* Children up to 14 years old;
* Written informed consent form signed by parents or legal guardians must be provided to caregivers.
* Subject willing and able to comply with study restrictions and willing to return to the health center and to perform the follow-up evaluation as specified in the protocol.

Exclusion Criteria:

* Use of antibiotics, diosmectite, probiotics, racecadotril, loperamide or zinc (including zinc containing ORS) within a week prior to enrolment
* Chronic diarrheal gastrointestinal disease (e.g, inflammatory bowel diseases, cystic fibrosis, coeliac disease, food allergy)
* Immunodeficiencies
* Signs of malnutrition according to the opinion of the investigator (weight/height under 3rd z score as per World Health Organization [WHO] Child Growth Standards)
* Need for Intravenous rehydration
* Subject who previously entered in a clinical study within the past 30 days.
* Pregnancy and suspected Pregnancy

Ages: 3 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhea | 48 hours
  Duration of diarrhea, defined as the time between start of diarrhea and the normalization of stool consistency according to the BSF or BITSS (in BSF scale, =3 or =4; in BITSS, =2), or/and the time until the normalization of the number of stools (compared with the period before the onset of diarrhea), and the presence of normal stools for 48 h.

CONTACTS AND LOCATIONS:
Overall Officials: Aldiouma Diallo, MS, Principal Investigator — IRD Senegal (Niakhar Center IRD BP 1386 Hann Mariste, CP 18524 Dakar. Sénégal.; Javier Xllop, Study Director — Noventure SL
Locations (1):
- Niakhar Center IRD, Dakar, Senegal